CLINICAL TRIAL: NCT04296071
Title: Neutrophil Phenotypic Profiling and Acute Lung Injury in Patients After Cardiopulmonary Bypass (CPB)
Status: Recruiting | Type: Observational
Sponsor: Sophia Koutsogiannaki (Other)
Responsible Party: Sponsor-Investigator, Sophia Koutsogiannaki, Assistant Professor, Boston Children's Hospital
Organization: Boston Children's Hospital (Other)
Other Study IDs: IRB-P00034280
Record Dates: First submitted 2020-03-03; First posted 2020-03-05 (Actual); Last update posted 2024-08-23 (Actual); Status verified 2024-08

CONDITIONS: Lung Injury; Cardiopulmonary Bypass
MeSH Terms: conditions — Lung Injury

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Samples Without DNA — Blood will be collected from existing intravenous or arterial catheters. Tracheal aspirates will be obtained by collecting the suction catheter used.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Group 1: patients who tend to have longer CPB
  Interventions: Other: Research study
- Group 2: Patients who have shorter CPB
  Interventions: Other: Research study

INTERVENTIONS:
Other: Research study — Blood and tracheal aspirates will be collected

SUMMARY:
Acute lung injury (ALI) following cardiopulmonary bypass (CPB) is a serious complication, often prolonging the length of stay in ICU and potentially dealing to mortality. The objective of this study is to assess the mechanism of CPB-mediated acute lung injury in pediatric patients.

DETAILED DESCRIPTION:
Acute lung injury (ALI) is frequently associated with the use of extracorporeal circulation during cardiopulmonary bypass (CPB) surgery and develops postoperatively in 2-3% of cardiac surgical patients. Histological evidence shows that CPB increases pulmonary vascular permeability and extravascular lung water content while diminishing pulmonary compliance. Furthermore, some patients can develop acute respiratory distress syndrome, which has a mortality rate of 50-70%. Recruitment of intrapulmonary neutrophils is a characteristic of ALI following CPB. Blood contact with non-physiological surfaces, cooling and rewarming and mechanical shear stress activate neutrophils. The recruitment of activated neutrophils from blood vessels to local tissue involves a chain of well-coordinated events, including adhesion, tethering, rolling and crawling, followed by trans-endothelial and trans-epithelial migration. Activation of sequestered neutrophils causes the release of specific proteolytic enzymes and oxygen free radicals, which leads to increased alveolar-endothelial permeability and parenchymal damage. During CPB, the lungs are almost completely excluded from the systemic circulation, which causes the blood within them to be almost 'static'. Pulmonary tissue hypoxia and re-oxygenation combined with vascular ischemia and reperfusion induce the generation of chemokines, which contributes to subsequent injury by accumulating and entrapping activated neutrophils. The accumuled and entrapped activated neutrophils in the lungs and the subsequent release of toxic substances render the lungs highly susceptible to this damage. However, the mechanism that drives neutrophil migration to the lungs after CPB is not well studied. This study will delineate the mechanisms of neutrophil migration to the lung and subsequent lung injury after CPB.

ELIGIBILITY:
Inclusion Criteria:

* Are < 12months of age
* Scheduled for cardiac surgical needing CPB
* Preoperative SpO2 > 90%

Exclusion Criteria:

* Lack of parental (or legal guardian's) consent
* Preoperative SpO2 < 90%
* Preoperative oxygen therapy

Max Age: 12 Months | Sex: All | Healthy Volunteers: No
Age Groups: Child
Study Population: We will enroll patients < 12 months of age who undergo CPB surgery. This patient population is associated with the highest incidence of morbidity and mortality following cardiac surgery, due to often prolonged period of CPB. Patients will be categorized into two groups: Group 1: patients who tend to have longer CPB (> 3 h), (ASO, Stage 1, IAA repair, Truncus repair, TAPVR) and Group 2: Patients who have shorter CPB (< 3hrs VSD, TOF, ASD).
Sampling Method: Non-Probability Sample
Enrollment: 56 (Estimated)
Dates: Start 2022-10-14 (Actual); Primary Completion 2026-04 (Estimated); Study Completion 2026-12 (Estimated)

PRIMARY OUTCOMES:
Perform neutrophil analysis in blood and tracheal aspirates samples | 2 years
  We will analyze neutrophil profiles in the blood and tracheal aspirates

SECONDARY OUTCOMES:
Determine chemoattractant levels | 2 years
  We will measure the levels of chemoattractants in the blood and tracheal aspirates
Determine neutrophil functions | 2 years
  We will measure neutrophil functions from the blood and tracheal aspirates

CONTACTS AND LOCATIONS:
Locations (1):
- Boston Children's Hospital, Boston, Massachusetts, United States

IPD SHARING:
Plan to Share IPD: No